CLINICAL TRIAL: NCT05316610
Title: Body Confident Athletes: Acceptability Testing of a Coach-Led Body Image Intervention for Adolescent Girls in Sport
Brief Title: Coach-Led Body Image Intervention for Girls in Sport - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); Nike (Industry); Laureus (Unknown); Tucker Center for Research on Girls & Women in Sport (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HAS.21.03.120a
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Intervention; Waitlist Control
Keywords: Body image; Embodiment; Girls; Athletes; Coaches; Task shifting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Confident Athletes (Experimental): Participants in the intervention condition will take part in an in-person program consisting of five sessions over five weeks.
  Interventions: Behavioral: Body Confident Athletes
- Waitlist control (No Intervention): Participants will not be explicitly told their study condition, although they will be made aware of the assessment time points and whether they receive the intervention between T1 and T2 (intervention) or after T2 (waitlist control). Following completion of post-intervention assessments (T2), the control condition will participate in the intervention; but, they will not be monitored or assessed.

INTERVENTIONS:
Behavioral: Body Confident Athletes — The Body Confident Athletes program is a five-session in-person program designed to be delivered by coaches to their athletes. Groups should be of approximately 10 girls. The organizations will work with the community partner and researchers on how to schedule the intervention over a five-week period. These sessions can replace a regular sport practice each week or an additional session can be organized by the sport organizations. Each session will take approximately 60 minutes and will consist of four phases, including The Game Plan (5 mins), The Skills (20 mins), Game Time (20 mins), and The Final Score (15 mins). A variety of activity modalities are utilized to convey learning outcomes, including group and individual activities, and discussion-, writing- and movement-based activities.
  Arms: Body Confident Athletes

SUMMARY:
According to the World Health Organization, only 15% of 11-17-year-old girls meet the recommended daily physical movement guidelines (e.g., 60-minutes per day). Despite extensive research highlighting the protective factors associated with sport on both mental and physical health, body image concerns are a key barrier to girls' participation in and enjoyment of sport. Sports-related environments and society more broadly further exacerbate these concerns through harmful gender stereotypes that perpetuate female objectification, discrimination, and harassment. This includes the promotion of unrealistic and sexualized appearances of female athletes, uncomfortable and objectifying uniforms, and appearance and competence-related teasing from male and female peers, as well as coaches.

The magnitude of this issue and how best to address it, can be understood from a socioecological perspective. Researchers suggest developing multi-faceted and multi-tiered approaches that have scope for targeting the individual, interpersonal, organizational, and societal levels. The current research will test the first coach delivered embodying sports program for girls that will be implemented through sporting organizations. The Body Confident Athletes program was co-created with girls and coaches through an international multi-disciplinary partnership between academics, health professionals, industry, and community organizations. Multi-disciplinary partnerships can create a supportive landscape by upskilling girls and influential community members (e.g., coaches) in dealing with body image concerns, which will likely lead to sustained sports participation and biopsychosocial benefits.

As such, the aim of the present study is to conduct a randomized controlled trial (RCT) to evaluate the effectiveness, feasibility, and acceptability of the Body Confident Athletes program. The program consists of five 60-minute sessions delivered by coaches to adolescent girls. Each session tackles a distinct theme related to body image in the sporting context. Outcomes will be assessed at pre- and post-intervention (5 weeks later) and include body image (primary outcome), sport enjoyment and embodied experiences (secondary outcomes), and feasibility, acceptability, and adherence (process outcomes). The comparison control arm will be a waitlist control condition.

To undertake this project, sporting organizations will be cluster-randomized into the intervention group or the control group, with 80 girls anticipated in each arm. Those in the intervention condition will complete baseline assessments (target outcomes and demographic information), take part in the five-week intervention, and then complete the post-intervention assessments (target outcomes and feasibility and acceptability measures). Those in the waitlist control condition will complete the baseline assessments (target outcomes and demographic information) and a second assessment five weeks later (target outcomes only), after which they will get access to the intervention. However, their engagement with the intervention will not be monitored or assessed. At completion of the post-intervention survey, all participants will receive a debrief form, outlining the study aims and objectives, and additional resources for body image and eating concerns. Lastly, to compensate participants for their time, girls and coaches will receive an electronic voucher to the value of $60 dollars.

The investigators hypothesize that girls who take part in the Body Confident Athletes intervention will report better body image, greater sport enjoyment, and higher levels of embodiment at post-intervention than girls who do not take part in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Girls aged 11-17 years old
* English speaking
* US resident

Exclusion Criteria:

* n/a

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in body esteem (assessed via the Body Esteem Scale for Adults and Adolescents) | Baseline, pre-intervention; immediately after the intervention (5 weeks later)
  The Body Esteem Scale for Adults and Adolescents (BESAA) assesses body esteem (BE), which refers to self-evaluations of one's body or appearance. The BESAA has 3 subscales: BE-Appearance (general feelings about appearance), BE-Weight (weight satisfaction), and BE-Attribution (evaluations attributed to others about one's body and appearance). BESAA scores range from 0-4 with higher scores on the BESAA indicating higher levels of body esteem.

SECONDARY OUTCOMES:
Change in embodiment (assessed via the Youth Experience of Embodiment Scale) | Baseline, pre-intervention; immediately after the intervention (5 weeks later)
  The Youth Experience of Embodiment Scale (YEES) assesses how girls inhabit their body (e.g., body connection and comfort, attuned self-care) and how they navigate the world (e.g., with agency, resisting self-objectification). YEES scores range from 1-5 with higher scores on the YEES indicating higher levels of embodiment.
Change in sport enjoyment (assessed via the Sources of Enjoyment in Youth Sport Questionnaire) | Baseline, pre-intervention; immediately after the intervention (5 weeks later)
  The Sources of Enjoyment in Youth Sport Questionnaire (SEYSQ) assesses the source of an athlete's enjoyment in sport according to two spectrums (intrinsic motivation vs. extrinsic motivation and achievement vs. non-achievement factors), resulting in four quadrants indicating the four sources of an athlete's enjoyment. SEYSQ scores range from 1-5.

OTHER OUTCOMES:
Total acceptability of the intervention (assessed via a self-report questionnaire) | Immediately after the intervention
  Girls and coaches will complete feasibility and acceptability measures via a self-report questionnaire. Firstly, girls and coaches will respond using a 1-5 scale (Strongly Disagree to Strongly Agree) on questions, such as: 1) The program was interesting; 2) The program was easy to understand; 3) The program was enjoyable; and 4) The program discussed things that are important to me. Secondly, girls and coaches will be able to provide further feedback using open-ended responses on questions such as: 1) What did you like about the program and why? 2) What would you change about the program and why? 3) What did you think about the design of the materials? 4) Please tell us anything else you think will help improve the program for girls.
Total intervention fidelity (assessed via investigator observation of recorded intervention sessions) | Immediately after the intervention
  Total intervention fidelity will be assessed by the investigators through observing the program sessions as delivered by coaches and completing a pre-determined checklist to ensure the program was delivered to girls as intended.
Total intervention adherence (assessed through session completion) | Immediately after the intervention
  Total intervention adherence will be assessed by the investigators as number of participants who complete the full intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Appearance Research, University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Global trends in insufficient physical activity among adolescents: a pooled analysis of 298 population-based surveys with 1.6 million participants. Lancet Child Adolesc Health. 2020 Jan;4(1):23-35. doi: 10.1016/S2352-4642(19)30323-2. Epub 2019 Nov 21. PMID 31761562
- [Background] Neumark-Sztainer D, MacLehose RF, Watts AW, Pacanowski CR, Eisenberg ME. Yoga and body image: Findings from a large population-based study of young adults. Body Image. 2018 Mar;24:69-75. doi: 10.1016/j.bodyim.2017.12.003. Epub 2017 Dec 27. PMID 29288970
- [Background] Sabiston, C., Pila, E., Vani, M., & Thogersen-Ntoumani, C. (2019). Body image, physical activity, and sport: A scoping review. Psychology Of Sport And Exercise, 42, 48-57. doi: 10.1016/j.psychsport.2018.12.010
- [Background] Sabiston, C. M., Vani, M. F., & Murray, R. M. (2021). Body-related self-conscious emotions in sport and exercise: A self-regulation perspective. In Motivation and Self-regulation in Sport and Exercise (pp. 62-77). Routledge.
- [Background] Slater A, Tiggemann M. Gender differences in adolescent sport participation, teasing, self-objectification and body image concerns. J Adolesc. 2011 Jun;34(3):455-63. doi: 10.1016/j.adolescence.2010.06.007. Epub 2010 Jul 31. PMID 20643477
- [Background] Vani MF, Pila E, Willson E, Sabiston CM. Body-related embarrassment: The overlooked self-conscious emotion. Body Image. 2020 Mar;32:14-23. doi: 10.1016/j.bodyim.2019.10.007. Epub 2019 Nov 13. PMID 31733410
- [Result] Matheson EL, Schneider J, Tinoco A, Gentili C, Silva-Breen H, LaVoi NM, White P, Diedrichs PC. The co-creation, initial piloting, and protocol for a cluster randomised controlled trial of a coach-led positive body image intervention for girls in sport. BMC Public Health. 2023 Jul 31;23(1):1467. doi: 10.1186/s12889-023-16360-w. PMID 37525161